CLINICAL TRIAL: NCT04698681
Title: Screening Protocol to Detect Mutation of KEAP1 or NRF2/NFE2L2 Genes in Patients With Stage IV, 1L Non-Small Cell Lung Cancer to Determine Eligibility for the KEAPSAKE Clinical Trial (NCT04265534)
Brief Title: NGS Screening Protocol to Detect Mutation of KEAP1 or NRF2/NFE2L2 Genes for the KEAPSAKE (CX-839-014) Trial
Status: Terminated | Type: Observational
Why Stopped: Lack of Clinical Benefit
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CX-839-016
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Non-Small Cell Lung Cancer; Non-squamous Non-small-cell Lung Cancer; Non-Squamous Non-Small Cell Neoplasm of Lung; KEAP1 Gene Mutation; NRF2 Mutation; NFE2L2 Gene Mutation
Keywords: NSCLC; KEAP1; NRF2; NFE2L2; LKB1; STK11; Next Generation Sequencing; NGS; Mutation; Gene; Pembrolizumab; Pemetrexed; Carboplatin; Placebo; Randomized; Chemotherapy; Immunotherapy; Targeted Therapy; Telaglenastat; Glutamine; Glutaminase; Glutathione; Front-line; First-line; Non-Squamous; Keytruda; Alimta; Guardant360 LDT; Liquid Biopsy; ctDNA; Biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma for NGS analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Biomarker Screening: Patients with stage IV nonsquamous NSCLC not previously treated with systemic therapy for metastatic disease and who meet all of study inclusion criteria and none of the exclusion criteria.

SUMMARY:
This is a multicenter screening protocol designed to identify patients with NSCLC who have tumor mutations in the KEAP1 or NRF2/NFE2L2 genes in order to determine potential eligibility for a biomarker selected clinical trial (CX-839-014, otherwise known as the KEAPSAKE trial). Circulating tumor DNA (ctDNA) present in blood samples collected from eligible patients will be analyzed by next generation sequencing (NGS) for selected biomarkers. A commercial liquid biopsy NGS test will be provided to study participants free of charge.

ELIGIBILITY:
Inclusion Criteria:

Patients with stage IV non-squamous non-small-cell lung cancer (NSCLC) who have not been previously treated with systemic therapy for metastatic disease, and meet all of the following:

1. Signed and dated NGS Informed Consent Form (ICF) by the patient (or legally acceptable representative (LAR), if applicable).
2. Biopsy-confirmed OR clinically suspected stage IV NSCLC not previously treated with systemic therapy for metastatic disease.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Age ≥ 18 years old on the day of signing informed consent.
5. Estimated life expectancy > 3 months.
6. At least one radiographically measurable lesion per RECIST v1.1 defined as a lesion that is ≥ 10 mm in longest diameter or lymph node that is ≥ 15 mm in short axis imaged by computed tomography (CT) scan or magnetic resonance imaging (MRI).
7. Clinically eligible to receive standard-of-care combination therapy with pemetrexed + carboplatin + Pembrolizumab (PCP) for stage IV disease.

Exclusion Criteria:

Any contraindication to pemetrexed, carboplatin, and Pembrolizumab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLS with Mutation of KEAP1 or NRF2/NFE2L2 Genes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Positive KEAP1 or NRF2/NFE2L2 mutational status, assessed by NGS of blood ctDNA | Up to 16 months
  The percentage of patients with nonsquamous NSCLC containing pathogenic NRF2/NFE2L2 and/or KEAP1 mutations

CONTACTS AND LOCATIONS:
Overall Officials: Emil Kuriakose, MD, Study Director — Calithera Biosciences, Inc
Locations (63):
- United States (63):
  - Southern Cancer Center, Daphne, Alabama
  - Southern Cancer Center - 3 Mobile Infirmary Circle, Mobile, Alabama
  - Southern Cancer Center - Dauphin St, Mobile, Alabama
  - Southern Cancer Center - Providence Hospital, Mobile, Alabama
  - Arizona Oncology Associates - Glendale, Glendale, Arizona
  - Arizona Oncology Associates - E. Highland Ave., Phoenix, Arizona
  - Arizona Oncology Associates - N. 27th Ave., Phoenix, Arizona
  - Arizona Oncology Associates, Scottsdale, Arizona
  - Arizona Oncology Associates - Tempe, Tempe, Arizona
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Rocky Mountain Cancer Centers - Colorado Springs, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers - Williams Street, Denver, Colorado
  - Rocky Mountain Cancer Centers - E. Hale Parkway, Denver, Colorado
  - Rocky Mountain Cancer Centers - Englewood, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers - Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers - Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Thornton, Thornton, Colorado
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Woodlands Medical Specialists, Pensacola, Florida
  - Maryland Oncology Hematology - Bethesda, Bethesda, Maryland
  - Maryland Oncology Hematology - Brandywine, Brandywine, Maryland
  - Maryland Oncology Hematology - Clinton, Clinton, Maryland
  - Maryland Oncology Hematology, Columbia, Maryland
  - Maryland Hematology Oncology - Frederick, Frederick, Maryland
  - Maryland Oncology Hematology - Lanham, Lanham, Maryland
  - Maryland Hematology Oncology - Rockville, Rockville, Maryland
  - Maryland Hematology Oncology - Silver Spring, Silver Spring, Maryland
  - Oncology Hematology Care - Mercy Health Blvd, Cincinnati, Ohio
  - Oncology Hematology Care - Malsbary Rd, Cincinnati, Ohio
  - Oncology Hematology Care - Ivy Gateway, Cincinnati, Ohio
  - Oncology Hematology Care - Fairfield, Fairfield, Ohio
  - Northwest Cancer Specialists - NE Hoyt St, Portland, Oregon
  - Northwest Cancer Specialists - N. Broadway, Portland, Oregon
  - Northwest Cancer Specialists, Tigard, Oregon
  - Consultants in Medical Oncology and Hematology, Broomall, Pennsylvania
  - Consultants in Medical Oncology and Hematology, Horsham, Pennsylvania
  - Consultants in Medical Oncology and Hematology, Wynnewood, Pennsylvania
  - Texas Oncology - West Texas Amarillo, Amarillo, Texas
  - Texas Oncology - Beaumont, Beaumont, Texas
  - Texas Oncology - Beaumont Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Carrollton, Carrollton, Texas
  - Texas Oncology - Denton, Denton, Texas
  - Texas Oncology - Flower Mound, Flower Mound, Texas
  - Texas Oncology Cancer Care and Research, Harlingen, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - West Texas Midland, Midland, Texas
  - Texas Oncology - West Texas Odessa, Odessa, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Weslaco, Weslaco, Texas
  - Texas Oncology - West Texas Wichita Falls, Wichita Falls, Texas
  - Virginia Oncology Associaties, Chesapeake, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Cancer Specialists, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington